CLINICAL TRIAL: NCT07001202
Title: Acceptability and Feasibility of a Preventive Indicated Intervention for Suicidality in University Students: Reframe-IT+U
Brief Title: Acceptability and Feasibility of Reframe-IT+U for Suicidality in University Students.
Acronym: Reframe-IT+U
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Jorge Gaete, Full Professor, Universidad de los Andes, Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FDI UAN23102 - Reframe-IT+U; FDI UAN23102 (Other: Ministerio de Educacion, Chile)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Suicidal Ideation; Depression Disorders; Anxiety
Keywords: Suicidal ideation prevention; Indicated prevention; Depression prevention; Anxiety prevention; University students; College students
MeSH Terms: conditions — Suicidal Ideation; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study pre and post.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reframe-IT+U (Experimental): The Reframe-IT+U program is an individualized preventive intervention based on cognitive behavioral therapy, with a problem-solving and help-seeking approach, delivered within the University with psychologists and supervision. The program consists of six weekly sessions of 60-90 minutes each.
  Interventions: Behavioral: Indicated Prevention for suicidality

INTERVENTIONS:
Behavioral: Indicated Prevention for suicidality — The Reframe-IT+U program is an individualized preventive intervention based on cognitive behavioral therapy, with a problem-solving and help-seeking approach, delivered within the University with psychologists and supervision. The program consists of six weekly sessions of 60-90 minutes each.

SUMMARY:
Mental health in university students is a growing concern worldwide. In Chile, previous studies have shown high rates of depressive symptoms, anxiety, and suicidal risk in this population. This study seeks to evaluate the acceptability and feasibility of a Cognitive Behavioral Therapy (CBT)-based intervention for the indicated prevention of suicidality in undergraduate students, and also to explore its impact on reducing suicidal ideation. A quasi-experimental before-and-after design will be used with a sample of students from the Universidad de los Andes who present mild to moderate suicidal risk. As this is a pilot study, a sample size calculation is not required, but we expect to recruit 20 subjects, which will allow us to conduct acceptability and feasibility assessments and collect data for a larger-scale study. A follow-up will consist of repeating the initial assessment questionnaire, which will be completed two and four months after the intervention. The methodology includes an initial interview to assess inclusion and exclusion criteria, signing informed consent, and developing a safety plan with the students. Following this, six weekly sessions (three in-person and three with digital components) of 60 minutes each will be held, focusing on emotional regulation, cognitive restructuring, and problem-solving. The intervention will be facilitated by trained psychologists, under the supervision of a trained psychologist or psychiatrist. To assess acceptability, the Client Satisfaction Questionnaire (CSQ-8) will be primarily used.

To assess outcomes, validated instruments will be applied, such as the Columbia Suicide Risk Scale (C-SSRS), the Patient Health Questionnaire-9 (PHQ-9) for depressive symptoms, the Generalized Anxiety Disorder 7 (GAD-7) for anxiety symptoms, the Short Form-12 Health Survey (SF-12) for quality of life, the Distress Tolerance Scale (DTS) for stress tolerance, the Community Assessment of Psychic Experiences-Positive (CAPE-P15) for psychotic symptoms, the Difficulties in Emotion Regulation Scale (DERS-E) for emotional regulation, the Social Problem-Solving Inventory-Revised (SPSI-R) for problem-solving, and the Cognitive-behavioural Therapy Skills Questionnaire (CBTSQ) for cognitive-behavioral skills. Reduction in suicidal ideation, satisfaction with the intervention, and program adherence will be measured.

The study hopes that the prevention program, along with the proposed assessments and procedures, will be appropriate and feasible in a university setting. This will allow progress toward a larger randomized controlled trial. Furthermore, it is expected that students in the intervention group will experience a reduction in suicidal ideation.

DETAILED DESCRIPTION:
Mental health among university students has become, in recent years, a common and serious issue within higher education institutions worldwide, and Chile is no exception.

A systematic review and meta-analysis published in 2022 found a global prevalence of depressive symptoms among university students of 33.6% and anxiety symptoms of 39%. In Latin America, a study conducted in Brazil (2017) among medical students showed a prevalence of depression of 30.6%, anxiety disorders of 32.9%, and stress of 49.9%.

In Chile, there are few studies addressing the prevalence of mental health disorders among university students. In the "First National University Mental Health Survey," conducted in 2018 among 600 students from the Catholic University of Temuco, the University of Concepción, and the University of Tarapacá, 46% of students showed depressive symptoms, 46% anxiety symptoms, and 53.5% stress symptoms. Additionally, 29.7% presented all three symptoms simultaneously, and 5.1% of students had suicidal thoughts.

Data from the first Mental Health Survey at Universidad de los Andes, conducted in 2020 with 5,037 undergraduate students, showed a prevalence of depressive symptoms of 37.1% and anxiety symptoms of 37.9%. The prevalence of suicide risk was 20.0%. In the second survey at this institution in 2022, with 1,682 students participating, the prevalence of depression was 27.84%, anxiety 36.12%, and stress 2.91%. Suicidal ideation risk was found to be 18.7%.

The prevalence of suicidal ideation is alarming. However, it aligns with information from the World Health Organization (WHO), which states that suicide is the second leading cause of death among youth aged 15 to 29 worldwide.

Recent literature regarding suicide among university students is concerning. In the updated study of the Ten Great Schools, published by the National Academies of Sciences, Engineering, and Medicine, researchers found a suicide mortality rate of 5.6 per 100,000 students between 2009 and 2018.

A meta-analysis including 634,662 university students found high proportions of students experiencing suicidal thoughts, plans, and behaviors. The pooled lifetime prevalence estimates of suicidal ideation, plans, and attempts were 22.3%, 6.1%, and 3.2%, respectively. For the past 12-month prevalence, these figures were 10.6%, 3.0%, and 1.2%, respectively.

A cross-sectional study conducted in 2023 with 12,245 university students in Brazil found a prevalence of suicidal ideation of 5.9%. Variables most associated with suicidal ideation included a history of psychopathology, sexual abuse, dissatisfaction with course choice, and low academic performance.

The above was presented as background for suicide risk, but suicidal behavior has also been shown to have significant consequences in university students' lives. Suicide attempts are the most significant risk factor for completed suicide. Suicidal ideation is also strongly associated with a greater risk of future suicide. Moreover, experiencing mental health problems is associated with poor academic performance and increased dropout rates, with a 210% increase in the number of students who dropped out of their studies due to mental health problems in the past four years.

A meta-analytic synthesis published in 2021 evaluated risk factors related to suicide among university students. Adverse childhood experiences, underlying mental health problems, and financial difficulties predicted a higher risk of suicidal ideation and behavior. Regarding sexual minorities, the American College Health Association (ACHA) reported that 5.4% of transgender and gender non-conforming university students had attempted suicide in the past year, compared to 2.9% of cisgender men and 1.9% of cisgender women.

Considering all of the above, mental health disorders among university students remain a public health issue that should be addressed preventively through the implementation of evidence-based programs.

Following a public health model, suicide prevention strategies can be implemented at three levels: universal, selective, and indicated. Universal interventions target the general population. Selective interventions focus on subpopulations at higher risk, which can be identified based on sociodemographic characteristics, geographic distribution, or prevalence of mental disorders and substance use. Finally, indicated interventions are aimed at individuals known to be vulnerable to suicide or who have previously attempted suicide. In the university population, indicated prevention targets students showing warning signs or identified with potential suicide risk. A comprehensive suicide prevention program typically employs a combination of universal, selective, and indicated interventions.

In the United Kingdom, there is a national suicide prevention strategy for university students called the Suicide Safer University Strategy. It is based on pre-training members of the university community to enable them to carry out prevention and intervention with students. As training programs, they recommend interactive one- or two-day workshops such as the Applied Suicide Intervention Skills Training (ASIST). In the United States, there is a student suicide prevention guide developed by the Suicide Prevention Center of New York State. The indicated prevention model focuses on assessment and triage using semi-structured interviews, risk level determination using instruments such as the Columbia scale, collaborative safety planning such as the Stanley-Brown Safety Plan, notifying the primary support network, and timely referral to community health providers.

In 2019, Chile published its first set of recommendations for suicide prevention in educational institutions, which consists of six pillars: creating and maintaining a protective climate, preventing mental health problems and disorders, educating and raising awareness about suicide, detecting students at risk, acting protocols in case of an attempt or suicide, and postvention actions, as well as coordination and access to the health network.

On the other hand, a successful mental health prevention program for university students should include strategies that promote emotion regulation, a crucial component of well-being and social adaptation. One of the psychological theories that has most contributed to the development of preventive and therapeutic interventions in emotion management is cognitive-behavioral theory. Likewise, the literature highlights the importance of developing skills to cope with academic stress, such as effective appraisal of stressful situations and the use of problem-solving strategies.

A systematic review of suicide prevention in schools and universities included 35 studies, with a total of 24,270 participants. Of those 35 studies, 15 correspond to indicated prevention, and only 6 interventions are for indicated prevention in university populations, with the rest conducted in school populations.

Among the included studies, Fitzpatrick et al. (2005) conducted a randomized controlled trial using a brief audiovisual intervention focused on problem-solving and coping strategies. They found a decrease in suicidal ideation and depression in the intervention group, although the difference was not significant compared to the control group (26% vs. 22% improvement; p > .10).

In a randomized controlled trial by Lin et al. (2019), a group of Taiwanese university students diagnosed with borderline personality disorder participated in a group cognitive-behavioral therapy (CBT) intervention aimed at reducing depression and suicide attempts. Another group participated in a skills training intervention based on dialectical behavior therapy (DBT). For the CBT group, a significant reduction in suicidal ideation was observed at 4, 8, 20, and 32 weeks of follow-up, with a large effect size (d = 5.24). For the DBT skills training group, a significant reduction in suicide attempts was found at 4, 8, 20, and 32 weeks of follow-up, with a small effect size (d = 0.32).

Instruments used to measure suicidal ideation and behavior included validated scales such as the Columbia Suicide Severity Rating Scale, the Beck Scale for Suicidal Ideation, and the Suicidal Behaviors Questionnaire-Revised (SBQ-R).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Undergraduate students at Universidad de los Andes.
* Able to read and speak Spanish.
* Mild to moderate suicide risk in the past month, defined as having answered "Yes" to items 1, 2, 3, and/or 4 on the Columbia Suicide Severity Rating Scale (C-SSRS).

Exclusion Criteria:

* Severe suicide risk, defined as having answered "Yes" to item 5 (past month) or item 6 (past 3 months) on the Columbia Suicide Severity Rating Scale (C-SSRS).
* Presence of a severe, untreated psychiatric condition during the past year or history of psychiatric hospitalization in the last two years.
* Determination by the University Wellness Team that the participant is not in a suitable condition to participate due to a severe psychiatric condition or need for hospitalization.
* High severity of psychotic symptoms (score equal to or greater than 2 on any of items 13, 14, and/or 15 of the Community Assessment of Psychic Experiences - Positive Scale (CAPE, P15)).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | End of intervention at 6 weeks
  It is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria from "0" (Never) to "3" (Almost Every Day). In Chile, it has been validated among people aged 20 years and over, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression Scale. In addition, it has construct validity and concurrent predictive validity with the The International Classification of Diseases, 10th Revision (CIE-10) criteria for depression. The interpretation is made by adding the total of the first nine questions: 0-4 points, without depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Feasibility Assessment: Number of participants recruited | through study completion, an average of 1 year
  Initially, inclusion and exclusion criteria will be defined to ensure that participants are representatives of the target group. A tracking system will be implemented to monitor the number of people recruited.
Feasibility Assessment: Recruitment time for completion | through study completion, an average of 1 year
  A tracking system will be implemented to monitor the time needed to complete the recruitment process.
Feasibility Assessment: Evaluation of data collection and results. | through study completion, an average of 1 year
  Clear protocols will be established for data collection and analysis, ensuring accuracy and consistency. Statistical analyzes will be used to check the validity and reliability of the results.
Feasibility Assessment: Level of progress of the participants in the sessions. | through study completion, an average of 1 yea
  The completion and the time needed for completion of each module of the intervention will be registered.

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (C-SSRS) | Through study completion, an average of 1 year
  The first 5 items explore the presence of suicidal ideation, intention, and planning and are assessed over the past month. The sixth item explores suicidal behavior either as preparation, initiation of a suicide attempt, or a suicide attempt itself in the last three months. Each item is answered Yes or No. It has been validated in an English-speaking population (range of internal reliability goes from α=0.73 to α=0.93) and a Spanish-speaking population (α=0.53). The total score range is from 0 to 6 points. According to the answers provided To the different items, the categories of severity of suicidal ideation are established: If the answer is "Yes" to item 1 and/or item 2 and "No" to all the other items, a slight risk is indicated. If the answer is "Yes" to item 2 and answer "Yes" only to item 3, it suggests that the risk is moderate. If the answer si "Yes" to item 2 and the answer is "Yes" to any of items 4, 5, and 6, it indicates that the risk is severe.
Patient Health Questionnaire-9 (PHQ-9) | Through study completion, an average of 1 year
  It is a self-administered version of the PRIME-MD diagnostic instrument for common mental disorders. The PHQ-9 is the depression module, which rates each of the 9 Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) criteria from "0" (Never) to "3" (Almost Every Day). In Chile, it has been validated among people aged 20 years and over, with a sensitivity of 92% and a specificity of 89%, compared to the Hamilton Depression Scale. In addition, it has construct validity and concurrent predictive validity with the The International Classification of Diseases, 10th Revision (CIE-10) criteria for depression. The interpretation is made by adding the total of the first nine questions: 0-4 points, without depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Generalized Anxiety Disorder (GAD-7) | Through study completion, an average of 1 year
  GAD-7 was originally designed primarily as a screening and severity measure for generalized anxiety disorder, this instrument also has good performance characteristics for other common anxiety disorders: panic disorder, social anxiety disorder, and post-traumatic stress disorder. This consists of 7 questions. The score is calculated by assigning scores from 0 to 3 to response categories from "Never" to "Almost Every Day." It has been validated in Spanish, where a cut-off score of 10 showed adequate values of sensitivity (86.8%) and specificity (93.4%). The scale was significantly correlated with Hamilton Anxiety scal (HAM-A) (0.852, p < 0.001), Hospital Anxiety and Depression Scale (HADS ) (anxiety domain, 0.903, p < 0.001), and World Health Organization Disability Scale (WHO-DAS II) (0.696, p < 0.001). The GAD-7 total score for the seven items ranges from 0 to 21
Distress Tolerance Scale (DTS) | Through study completion, an average of 1 year
  This instrument allows us to evaluate how people experience and endure distressing psychological states. The scale is constructed of 15 items, divided into four subscales that measure four factors: Tolerance (items 1, 3, and 5), understood as the perceived ability to handle strong emotions; Relief (items 2, 4, and 15), considered as "how relieved a person feels when they experience a strong emotion"; Evaluation (items 6, 7, 9, 10, 11 and 12), understood as the person's perceived ability to accept their strong emotions; and, Regulation (items 8, 13 and 14), understood as the effort that a person makes to manage their intense emotions openly. DTS is a scale designed to be self-administered that is answered using a type format.
The Cognitive-behavioral Therapy Skills Questionnaire (CBTSQ) | Through study completion, an average of 1 year
  Evaluates which components of Cognitive behavioral therapy (CBT) appear to be most active. This scale originally has 16 items that measures two skills: cognitive restructuring (CR) and behavioral activation (BA). Respondents rate each item on a 5-point Likert scale, from 1 (I don't do this) to 5 (I always do this). Both scales have good reliability (CR: α=0.88; BA: α=0.85). Two items refer to evaluating aspects related to a disease or treatment. Since cognitive-behavioral skills are evaluated in this study, these two items of the questionnaire are included, leaving an instrument of 14 items. In a study whose publication is under review with adolescents between 15 and 18 years old, using the 14-item instrument, it was found that the reliability was α=0.77 and ω=0.78 for BA and α=0, 80 and ω=0.81 for CR. The minimum score would be 14 and the maximum would be 70. A higher score on the CBTSQ indicates greater competence and use of cognitive behavioral therapy skills.
Community Assessment of Psychotic Experiences Scale (CAPE-P15) | Through study completion, an average of 1 year
  This is a 15-item self-report instrument. Item responses range from 1 (never) to 5 (very often). The scale assesses three domains: paranoid ideation (PI, 5 items), bizarre experiences (EB, 7 items), and perceptual anomalies (AP, 3 items). Scores can range from 15 to 75. Higher scores indicate greater severity of Psychotic Experiences. All items are averaged for an overall measure of the trait being assessed. In a validation study of a Chilean population of adolescents between 13 and 18 years of age, the trifactorial nature of the scale was confirmed. Internal reliability for these factors was 0.779 for PI; 0.839 for EB; and 0.884 for AP.
Brief Problem Solving Inventory (SPSI-R) | Through study completion, an average of 1 year
  This is a 25-item self-report instrument that measures two adaptive problem-solving dimensions (positive problem orientation and rational problem solving) and three dysfunctional dimensions (negative problem orientation, impulsive/careless style, and avoidant style). Each item is rated on a 5-point scale ranging from not at all true for me (0) to extremely true for me (4). The Spanish version has the same factor structure and appropriate alpha coefficients for the five subscales (from 0.62 to 0.99), and an overall internal consistency of 0.90 in Chilean adolescents. In our sample at baseline, Cronbach's α was 0.83 and McDonald's ω was 0.83 on an overall scale.
Difficulties in Emotion Regulation Scale - Spanish Version (DERS-E) | Through study completion, an average of 1 year
  The DERS-E is a self-report questionnaire designed to assess difficulties in emotion regulation. This instrument measures variables such as emotional dyscontrol, daily life interference, emotional inattention, emotional confusion, and emotional rejection. The Spanish-adapted version of the DERS, originally developed by Gratz and Roemer (2004), contains 28 items distributed across five subscales, compared to the original version's 36 items and six subscales. Items are rated using a five-point Likert scale (1 = almost never, 5 = almost always), where higher scores indicate greater difficulties in emotion regulation. The psychometric properties of the DERS-E show adequate internal consistency with Cronbach's alpha ranging from = 0.71 to 0.73, and good test-retest reliability over a six-month period (ρ = 0.74, p < 0.001).
12-item Short-Form Health Survey | Through study completion, an average of 1 year
  The SF-12 is an instrument that assesses quality of life and general health status. It consists of twelve items aimed at evaluating the level of well-being and functional capacity in individuals over 14 years old, defining both positive and negative states of physical and mental health through eight dimensions (physical functioning, physical role, bodily pain, mental health, general health, vitality, social functioning, and emotional role). Response options follow a Likert-type scale (with the number of options ranging from three to six points, depending on the item), which assess the intensity and/or frequency of the person's health status. Scores range from 0 to 100, with higher scores indicating better health-related quality of life. Research using the twelve SF items has shown that this instrument is a valid and reliable measure, with internal consistency estimates above 0.70 and significant correlations. In the Chilean validation with an adult population, internal consistency was

IPD SHARING:
Plan to Share IPD: No
The data collected during the current study will be available from the Principal Investigator on reasonable request, with anonymized data.

REFERENCES:
- [Background] Ramirez S., Romo V., Gaete J. Prevalencia de Problemas de Salud Mental en los Estudiantes de Pregrado de la Universidad de los Andes. Santiago, Chile.: Centro de Investigación en Salud Mental Estudiantil. Universidad de los Andes; 2023.)
- [Background] Martínez, P., Jiménez-Molina, Á., Mac-Ginty, S., Martínez, V., & Rojas, G. (2021). Salud mental en estudiantes de educación superior en Chile: Una revisión de alcance con meta-análisis. Terapia Psicológica, 39(3), 405-423. http://dx.doi.org/10.4067/S0718-48082021000300405
- [Result] Valdes JM, Diaz FJ, Christiansen PM, Lorca GA, Solorza FJ, Alvear M, Ramirez S, Nunez D, Araya R, Gaete J. Mental Health and Related Factors Among Undergraduate Students During SARS-CoV-2 Pandemic: A Cross-Sectional Study. Front Psychiatry. 2022 May 31;13:833263. doi: 10.3389/fpsyt.2022.833263. eCollection 2022. PMID 35711588
- [Result] Li W, Zhao Z, Chen D, Peng Y, Lu Z. Prevalence and associated factors of depression and anxiety symptoms among college students: a systematic review and meta-analysis. J Child Psychol Psychiatry. 2022 Nov;63(11):1222-1230. doi: 10.1111/jcpp.13606. Epub 2022 Mar 16. PMID 35297041
- [Result] Pacheco JP, Giacomin HT, Tam WW, Ribeiro TB, Arab C, Bezerra IM, Pinasco GC. Mental health problems among medical students in Brazil: a systematic review and meta-analysis. Braz J Psychiatry. 2017 Oct-Dec;39(4):369-378. doi: 10.1590/1516-4446-2017-2223. Epub 2017 Aug 31. PMID 28876408
- [Result] Mortier P, Cuijpers P, Kiekens G, Auerbach RP, Demyttenaere K, Green JG, Kessler RC, Nock MK, Bruffaerts R. The prevalence of suicidal thoughts and behaviours among college students: a meta-analysis. Psychol Med. 2018 Mar;48(4):554-565. doi: 10.1017/S0033291717002215. Epub 2017 Aug 14. PMID 28805169
- [Result] Altavini CS, Asciutti APR, Santana GL, Solis ACO, Andrade LH, Oliveira LG, Andrade AG, Gorenstein C, Wang YP. Suicide ideation among Brazilian college students: Relationship with academic factors, mental health, and sexual abuse. J Affect Disord. 2023 May 15;329:324-334. doi: 10.1016/j.jad.2023.02.112. Epub 2023 Feb 26. PMID 36849006
- [Result] Brown GK, Beck AT, Steer RA, Grisham JR. Risk factors for suicide in psychiatric outpatients: a 20-year prospective study. J Consult Clin Psychol. 2000 Jun;68(3):371-7. PMID 10883553
- [Result] Joiner TE Jr, Brown JS, Wingate LR. The psychology and neurobiology of suicidal behavior. Annu Rev Psychol. 2005;56:287-314. doi: 10.1146/annurev.psych.56.091103.070320. PMID 15709937
- [Result] Hysenbegasi A, Hass SL, Rowland CR. The impact of depression on the academic productivity of university students. J Ment Health Policy Econ. 2005 Sep;8(3):145-51. PMID 16278502
- [Result] Megivern D, Pellerito S, Mowbray C. Barriers to higher education for individuals with psychiatric disabilities. Psychiatr Rehabil J. 2003 Winter;26(3):217-31. doi: 10.2975/26.2003.217.231. PMID 12653444
- [Result] Sheldon E, Simmonds-Buckley M, Bone C, Mascarenhas T, Chan N, Wincott M, Gleeson H, Sow K, Hind D, Barkham M. Prevalence and risk factors for mental health problems in university undergraduate students: A systematic review with meta-analysis. J Affect Disord. 2021 May 15;287:282-292. doi: 10.1016/j.jad.2021.03.054. Epub 2021 Mar 26. PMID 33812241
- [Result] Gould MS, Cross W, Pisani AR, Munfakh JL, Kleinman M. Impact of Applied Suicide Intervention Skills Training on the National Suicide Prevention Lifeline. Suicide Life Threat Behav. 2013 Dec;43(6):676-91. doi: 10.1111/sltb.12049. Epub 2013 Jul 25. Erratum In: Suicide Life Threat Behav. 2015 Apr;45(2):260. PMID 23889494
- [Result] Haeuser E, Serfes AL, Cork MA, Yang M, Abbastabar H, Abhilash ES, Adabi M, Adebayo OM, Adekanmbi V, Adeyinka DA, Afzal S, Ahinkorah BO, Ahmadi K, Ahmed MB, Akalu Y, Akinyemi RO, Akunna CJ, Alahdab F, Alanezi FM, Alanzi TM, Alene KA, Alhassan RK, Alipour V, Almasi-Hashiani A, Alvis-Guzman N, Ameyaw EK, Amini S, Amugsi DA, Ancuceanu R, Anvari D, Appiah SCY, Arabloo J, Aremu O, Asemahagn MA, Jafarabadi MA, Awedew AF, Quintanilla BPA, Ayanore MA, Aynalem YA, Azari S, Azene ZN, Darshan BB, Babalola TK, Baig AA, Banach M, Barnighausen TW, Bell AW, Bhagavathula AS, Bhardwaj N, Bhardwaj P, Bhattacharyya K, Bijani A, Bitew ZW, Bohlouli S, Bolarinwa OA, Boloor A, Bozicevic I, Butt ZA, Cardenas R, Carvalho F, Charan J, Chattu VK, Chowdhury MAK, Chu DT, Cowden RG, Dahlawi SMA, Damiani G, Darteh EKM, Darwesh AM, das Neves J, Weaver ND, De Leo D, De Neve JW, Deribe K, Deuba K, Dharmaratne S, Dianatinasab M, Diaz D, Didarloo A, Djalalinia S, Dorostkar F, Dubljanin E, Duko B, El Tantawi M, El-Jaafary SI, Eshrati B, Eskandarieh S, Eyawo O, Ezeonwumelu IJ, Ezzikouri S, Farzadfar F, Fattahi N, Fauk NK, Fernandes E, Filip I, Fischer F, Foigt NA, Foroutan M, Fukumoto T, Gad MM, Gaidhane AM, Gebregiorgis BG, Gebremedhin KB, Getacher L, Ghadiri K, Ghashghaee A, Golechha M, Gubari MIM, Gugnani HC, Guimaraes RA, Haider MR, Haj-Mirzaian A, Hamidi S, Hashi A, Hassanipour S, Hassankhani H, Hayat K, Herteliu C, Ho HC, Holla R, Hosseini M, Hosseinzadeh M, Hwang BF, Ibitoye SE, Ilesanmi OS, Ilic IM, Ilic MD, Islam RM, Iwu CCD, Jakovljevic M, Jha RP, Ji JS, Johnson KB, Joseph N, Joshua V, Joukar F, Jozwiak JJ, Kalankesh LR, Kalhor R, Kamyari N, Kanchan T, Matin BK, Karimi SE, Kayode GA, Karyani AK, Keramati M, Khan EA, Khan G, Khan MN, Khatab K, Khubchandani J, Kim YJ, Kisa A, Kisa S, Kopec JA, Kosen S, Laxminarayana SLK, Koyanagi A, Krishan K, Defo BK, Kugbey N, Kulkarni V, Kumar M, Kumar N, Kusuma D, La Vecchia C, Lal DK, Landires I, Larson HJ, Lasrado S, Lee PH, Li S, Liu X, Maleki A, Malik P, Mansournia MA, Martins-Melo FR, Mendoza W, Menezes RG, Mengesha EW, Meretoja TJ, Mestrovic T, Mirica A, Moazen B, Mohamad O, Mohammad Y, Mohammadian-Hafshejani A, Mohammadpourhodki R, Mohammed S, Mohammed S, Mokdad AH, Moradi M, Moraga P, Mubarik S, Mulu GBB, Mwanri L, Nagarajan AJ, Naimzada MD, Naveed M, Nazari J, Ndejjo R, Negoi I, Ngalesoni FN, Nguefack-Tsague G, Ngunjiri JW, Nguyen CT, Nguyen HLT, Nnaji CA, Noubiap JJ, Nunez-Samudio V, Nwatah VE, Oancea B, Odukoya OO, Olagunju AT, Olakunde BO, Olusanya BO, Olusanya JO, Bali AO, Onwujekwe OE, Orisakwe OE, Otstavnov N, Otstavnov SS, Owolabi MO, Mahesh PA, Padubidri JR, Pana A, Pandey A, Pandi-Perumal SR, Kan FP, Patton GC, Pawar S, Peprah EK, Postma MJ, Preotescu L, Syed ZQ, Rabiee N, Radfar A, Rafiei A, Rahim F, Rahimi-Movaghar V, Rahmani AM, Ramezanzadeh K, Rana J, Ranabhat CL, Rao SJ, Rawaf DL, Rawaf S, Rawassizadeh R, Regassa LD, Rezaei N, Rezapour A, Riaz MA, Ribeiro AI, Ross JM, Rubagotti E, Rumisha SF, Rwegerera GM, Moghaddam SS, Sagar R, Sahiledengle B, Sahu M, Salem MR, Kafil HS, Samy AM, Sartorius B, Sathian B, Seidu AA, Shaheen AA, Shaikh MA, Shamsizadeh M, Shiferaw WS, Shin JI, Shrestha R, Singh JA, Skryabin VY, Skryabina AA, Soltani S, Sufiyan MB, Tabuchi T, Tadesse EG, Taveira N, Tesfay FH, Thapar R, Tovani-Palone MR, Tsegaye GW, Umeokonkwo CD, Unnikrishnan B, Villafane JH, Violante FS, Vo B, Vu GT, Wado YD, Waheed Y, Wamai RG, Wang Y, Ward P, Wickramasinghe ND, Wilson K, Yaya S, Yip P, Yonemoto N, Yu C, Zastrozhin MS, Zhang Y, Zhang ZJ, Hay SI, Dwyer-Lindgren L; Local Burden of Disease sub-Saharan Africa HIV Prevalence Collaborators. Mapping age- and sex-specific HIV prevalence in adults in sub-Saharan Africa, 2000-2018. BMC Med. 2022 Dec 19;20(1):488. doi: 10.1186/s12916-022-02639-z. PMID 36529768
- [Result] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Result] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Result] Murphy MJ, Newby JM, Butow P, Loughnan SA, Joubert AE, Kirsten L, Allison K, Shaw J, Shepherd HL, Smith J, Andrews G. Randomised controlled trial of internet-delivered cognitive behaviour therapy for clinical depression and/or anxiety in cancer survivors (iCanADAPT Early). Psychooncology. 2020 Jan;29(1):76-85. doi: 10.1002/pon.5267. Epub 2019 Nov 12. PMID 31659822
- [Result] Breet E, Matooane M, Tomlinson M, Bantjes J. Systematic review and narrative synthesis of suicide prevention in high-schools and universities: a research agenda for evidence-based practice. BMC Public Health. 2021 Jun 10;21(1):1116. doi: 10.1186/s12889-021-11124-w. PMID 34112141
- [Result] Lin TJ, Ko HC, Wu JY, Oei TP, Lane HY, Chen CH. The Effectiveness of Dialectical Behavior Therapy Skills Training Group vs. Cognitive Therapy Group on Reducing Depression and Suicide Attempts for Borderline Personality Disorder in Taiwan. Arch Suicide Res. 2019 Jan-Mar;23(1):82-99. doi: 10.1080/13811118.2018.1436104. Epub 2018 May 10. PMID 29528807
- [Result] Beck AT, Kovacs M, Weissman A. Assessment of suicidal intention: the Scale for Suicide Ideation. J Consult Clin Psychol. 1979 Apr;47(2):343-52. doi: 10.1037//0022-006x.47.2.343. No abstract available. PMID 469082
- [Result] McMain SF, Guimond T, Barnhart R, Habinski L, Streiner DL. A randomized trial of brief dialectical behaviour therapy skills training in suicidal patients suffering from borderline disorder. Acta Psychiatr Scand. 2017 Feb;135(2):138-148. doi: 10.1111/acps.12664. Epub 2016 Nov 13. PMID 27858962
- [Result] Nunez D, Meza D, Andaur J, Robinson J, Gaete J. Reframe-IT+, an indicated preventive school-based intervention, reduces suicidal ideation among adolescents in vulnerable contexts in Chile. BMC Psychol. 2024 Dec 24;12(1):780. doi: 10.1186/s40359-024-02300-9. PMID 39719648
- [Result] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Result] Crockett MA, Martinez V, Ordonez-Carrasco JL. [Psychometric properties of the Generalized Anxiety Disorder 7-item (GAD-7) scale in Chilean adolescents]. Rev Med Chil. 2022 Apr;150(4):458-464. doi: 10.4067/S0034-98872022000400458. Spanish. PMID 36155755
- [Result] Garcia-Campayo J, Zamorano E, Ruiz MA, Pardo A, Perez-Paramo M, Lopez-Gomez V, Freire O, Rejas J. Cultural adaptation into Spanish of the generalized anxiety disorder-7 (GAD-7) scale as a screening tool. Health Qual Life Outcomes. 2010 Jan 20;8:8. doi: 10.1186/1477-7525-8-8. PMID 20089179
- [Result] Argyropoulos SV, Ploubidis GB, Wright TS, Palm ME, Hood SD, Nash JR, Taylor AC, Forshall SW, Anderson IM, Nutt DJ, Potokar JP. Development and validation of the Generalized Anxiety Disorder Inventory (GADI). J Psychopharmacol. 2007 Mar;21(2):145-52. doi: 10.1177/0269881107069944. PMID 17329293
- [Result] Andrews G. A brief integer scorer for the SF-12: validity of the brief scorer in Australian community and clinic settings. Aust N Z J Public Health. 2002 Dec;26(6):508-10. doi: 10.1111/j.1467-842x.2002.tb00357.x. PMID 12530792
- [Result] Lera L, Marquez C, Saguez R, Moya MO, Angel B, Albala C. [Quality of life of older people with depression and dependence: validity of the SF-12 (short form health survey) questionnaire]. Rev Med Chil. 2021 Sep;149(9):1292-1301. doi: 10.4067/S0034-98872021000901292. Spanish. PMID 35319682
- [Result] Sandin B, Simons JS, Valiente RM, Simons RM, Chorot P. Psychometric properties of the spanish version of The Distress Tolerance Scale and its relationship with personality and psychopathological symptoms. Psicothema. 2017 Aug;29(3):421-428. doi: 10.7334/psicothema2016.239. PMID 28693717
- [Result] Capra C, Kavanagh DJ, Hides L, Scott JG. Current CAPE-15: a measure of recent psychotic-like experiences and associated distress. Early Interv Psychiatry. 2017 Oct;11(5):411-417. doi: 10.1111/eip.12245. Epub 2015 May 12. PMID 25962504
- [Result] Nunez D, Arias V, Vogel E, Gomez L. Internal structure of the Community Assessment of Psychic Experiences-Positive (CAPE-P15) scale: Evidence for a general factor. Schizophr Res. 2015 Jul;165(2-3):236-42. doi: 10.1016/j.schres.2015.04.018. Epub 2015 Apr 30. PMID 25935814
- [Result] D'Zurilla TJ, Chang EC, Nottingham EJ 4th, Faccini L. Social problem-solving deficits and hopelessness, depression, and suicidal risk in college students and psychiatric inpatients. J Clin Psychol. 1998 Dec;54(8):1091-107. doi: 10.1002/(sici)1097-4679(199812)54:83.0.co;2-j. PMID 9840781
- [Result] De La Torre MT, Morera OF, Wood JM. Measuring social problem solving using the Spanish version for Hispanics of the Social Problem Solving Inventory-Revised. Cultur Divers Ethnic Minor Psychol. 2010 Oct;16(4):501-6. doi: 10.1037/a0021372. PMID 21058813
- [Result] Crockett MA, Martinez V, Jimenez-Molina A. Subthreshold depression in adolescence: Gender differences in prevalence, clinical features, and associated factors. J Affect Disord. 2020 Jul 1;272:269-276. doi: 10.1016/j.jad.2020.03.111. Epub 2020 Apr 29. PMID 32553367
- [Result] Jacob KL, Christopher MS, Neuhaus EC. Development and validation of the cognitive-behavioral therapy skills questionnaire. Behav Modif. 2011 Nov;35(6):595-618. doi: 10.1177/0145445511419254. Epub 2011 Sep 5. PMID 21893554
- [Result] Attkisson CC, Zwick R. The client satisfaction questionnaire. Psychometric properties and correlations with service utilization and psychotherapy outcome. Eval Program Plann. 1982;5(3):233-7. doi: 10.1016/0149-7189(82)90074-x. PMID 10259963
- [Result] Roberts RE, Attkisson CC. Assessing client satisfaction among Hispanics. Eval Program Plann. 1983;6(3-4):401-13. doi: 10.1016/0149-7189(83)90019-8. PMID 10267267
- [Derived] Gaete J, Nunez D, Romo V, Meza D, Robinson J, Araya R. Acceptability and feasibility of Reframe-IT+U for suicidal ideation in university students: protocol of a quasi-experimental pilot study. Pilot Feasibility Stud. 2025 Dec 8;12(1):7. doi: 10.1186/s40814-025-01738-x. PMID 41361289